CLINICAL TRIAL: NCT03600844
Title: Evaluation of Community Delivery of Malaria Intermittent Preventive Treatment in Pregnancy (C-IPTp) (TIPTOP Project)
Brief Title: Evaluating the Effects of Community Delivery of Malaria Intermittent Preventive Treatment on Pregnant Women and Babies
Acronym: TIPTOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jhpiego (Other)
Collaborators: Barcelona Institute for Global Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TIPTOP_HHS_2018; 2017-13-TIPTOP (Other Grant/Funding Number: Unitaid)
Record Dates: First submitted 2018-06-22; First posted 2018-07-26 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Malaria in Pregnancy

STUDY DESIGN:
Intervention Model Description: Districts in high malaria transmission zones were assigned to intervention and comparison areas.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phase 1 Intervention (Experimental): Phase 1 intervention communities will be offered Community distribution of SP for IPTp in addition to routine ANC IPTp distribution throughout the project.
  Interventions: Behavioral: Community distribution of SP for IPTp
- Phase 1 Comparison/Phase 2 Intervention (Active Comparator): During Phase 1 (intervention months 1 through 12), these communities will be offered only usual treatment--SP for IPTp at in facilities during routine ANC. During Phase 2 (intervention month 13 through the end of the project), these communities will be offered Community distribution of SP for IPTp, in addition to routine ANC IPTp distribution.
  Interventions: Behavioral: Community distribution of SP for IPTp

INTERVENTIONS:
Behavioral: Community distribution of SP for IPTp — SP is distributed to eligible pregnant women by trained Community Health Workers (CHWs) at community level. Demand creation activities are implemented within the community as well.
  Other Names: C-IPTp-SP

SUMMARY:
This study evaluates the effectiveness of community delivery of sulfadoxine-pyrimetamine (SP) for intermittent preventive treatment of malaria in pregnancy (IPTp) in increasing the coverage of IPTp among pregnant women in selected districts in Democratic Republic of Congo (DRC), Madagascar, Mozambique and Nigeria, compared to comparison districts where SP for IPTp is distributed as usual in facilities through routine antenatal care (ANC).

DETAILED DESCRIPTION:
The specific objectives of this study are to determine the change in the following indicators during the course of the TIPTOP project: 1) Proportion of women who have had a pregnancy that ended in the past 12 months and have received 1 or more, 2 or more and 3 or more doses of IPTp-SP; proportion of women with pregnancy in the past 12 months who attended ANC clinics at least once, and who attended at least four times; proportion of pregnant women attending the first ANC visit before or at week 14; proportion of women who have had a pregnancy that ended in the past 12 months who know about the IPTp service provided by CHWs; and acceptability of C-IPTp for community delivery of IPTp (note: results will be disaggregated by provider type, age, gravidity and distance from facility). To assess these changes, the study will implement structured household surveys targeting potential beneficiaries of the project (pregnant women) in the intervention and comparison areas, implemented at three time points: baseline, mid- and end-points. In each country an initial implementation area (Phase I) and two expansion areas (Phase II) have been selected for the project. This study will establish if community deliver of IPTp is effective and feasible and whether it influences antenatal care service coverage rates. It is expected that the study will provide information to scale up the approach the 4 study countries for the prevention of malaria in pregnancy. This information is also meant to inform global guidelines on community IPTp delivery and may also be used by other countries.

ELIGIBILITY:
Inclusion Criteria:

* Women who had a pregnancy that ended in the 12 months preceding the survey
* Being resident in the study area during for at least 4 months before the end of the pregnancy
* Willing to participate in the household survey (signing informed consent/assent, in line with country guidelines)

Exclusion Criteria:

* Anyone considered to be a minor in their country.
* Not willing to provide informed consent

Ages: 15 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 10602 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
IPTp3 Coverage | 1 year
  Proportion of women who had a pregnancy ending in the past 12 months and have received three or more doses of IPTp-SP

SECONDARY OUTCOMES:
IPTp1 Coverage | 1 year
  Proportion of women who have had a pregnancy that ended in the past 12 months and have received one or more doses of IPTp-SP
ANC 4 coverage | 1 year
  • Proportion of women who have had a pregnancy that ended in the past 12 months and have attended ANC clinics four times
ANC 1 Coverage | 1 year
  Proportion of women who have had a pregnancy that ended in the past 12 months and have attended ANC clinics at least once
Early ANC Coverage | 1 year
  Proportion of pregnant women attending the first ANC visit before or at week 14
C-IPTp Knowledge | 1 year
  Proportion of women who have had a pregnancy that ended in the past 12 months who know about the IPTp service provided by CHWs

CONTACTS AND LOCATIONS:
Overall Officials: Clara Menendez, MD, PhD, Principal Investigator — Barcelona Institute for Global Health
Locations (12):
- Democratic Republic of the Congo (3):
  - Kenge District, Community Setting, Kenge, Kwango
  - Bulungu District, Community Setting, Bulungu, Kwilu
  - Community Setting, Kunda, Maniema Province
- Madagascar (3):
  - Mananjary District, Community Setting, Mananjary, Fianarantsoa
  - Community Setting, Toliara, Fianarantsoa
  - Community Setting, Vohipeno, Vatovavy-Fitovinany
- Mozambique (3):
  - Meconta District, Community Setting, Meconta, Nampula
  - Community Setting, Murrupula, Nampula
  - Nhamatanda District, Community Setting, Nhamatanda, Sofala
- Nigeria (3):
  - Community Setting, Ohaukwu District, Ebonyi State
  - Community Setting, Bosso, Niger State
  - Community Setting, Akure South, Ondo State

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD to other researchers

REFERENCES:
- [Derived] Gonzalez R, Manun'Ebo MF, Meremikwu M, Rabeza VR, Sacoor C, Figueroa-Romero A, Arikpo I, Macete E, Mbombo Ndombe D, Ramananjato R, LIach M, Pons-Duran C, Sanz S, Ramirez M, Cirera L, Maly C, Roman E, Pagnoni F, Menendez C. The impact of community delivery of intermittent preventive treatment of malaria in pregnancy on its coverage in four sub-Saharan African countries (Democratic Republic of the Congo, Madagascar, Mozambique, and Nigeria): a quasi-experimental multicentre evaluation. Lancet Glob Health. 2023 Apr;11(4):e566-e574. doi: 10.1016/S2214-109X(23)00051-7. PMID 36925177
- [Derived] Pons-Duran C, Llach M, Sanz S, Ramirez M, Mendez S, Roman E, Tholandi M, Pagnoni F, Menendez C, Gonzalez R. Community delivery of malaria intermittent preventive treatment in pregnancy: protocol of a quasi-experimental evaluation through multistage cluster sampling household surveys in four sub-Saharan African countries. BMJ Open. 2021 Mar 25;11(3):e044680. doi: 10.1136/bmjopen-2020-044680. PMID 33766844